CLINICAL TRIAL: NCT06970028
Title: Somatosensory Phenotyping of Patients With ADPKD Using Quantitative Sensory Testing and Questionnaires
Brief Title: Somatosensory Phenotyping of ADPKD
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S70540
Record Dates: First submitted 2025-04-15; First posted 2025-05-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-04

CONDITIONS: ADPKD; Pain
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Pain | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ADPKD: Patients with ADPKD will be included (≥ 12 years old). The somatosensory profile will be described using Quantitative Sensory Testing and questionnaires regarding pain and quality of life.
  Interventions: Other: Quantitative Sensory Testing; Other: Questionnaires regarding pain and quality of life
- Healthy volunteers: Healthy volunteers will be included (≥ 12 years old), matched with the patient group based on age, sex and BMI. The somatosensory profile will be described using Quantitative Sensory Testing and the BPI-SF questionnaire.
  Interventions: Other: Quantitative Sensory Testing

INTERVENTIONS:
Other: Quantitative Sensory Testing — We will perform QST on the dominant hand and lower back.
Other: Questionnaires regarding pain and quality of life — Questionnaires will be filled out by patients with ADPKD to evaluate pain and quality of life.
  Groups: Patients with ADPKD

SUMMARY:
Over 60% of patients with ADPKD suffer from pain, mostly in the abdomen, flank and back, often leading to the diagnosis. It is challenging to manage and cure the pain; approximately 39% of patients are not satisfied with their pain treatment, since the pain prevents them from doing various activities, affecting their quality of life. Pain can be present before enlargement of the kidneys, the source of the pain is often unknown and common analgesics are insufficient to manage the pain or cannot be taken due to renal impairment. By further investigating and characterizing the pain phenotype of the ADPKD population, pain management might be improved and alternative therapeutic approaches might be developed. In this clinical study, pain will be assessed in patients with ADPKD using Quantitative Sensory Testing (QST) on the dominant hand and the lower back, together with four questionnaires regarding pain and quality of life. These results will be compared with the somatosensory profile of matched healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Patients with ADPKD

* Subject is ≥ 12 years old.
* Subject is diagnosed with ADPKD.

Healthy volunteers

* Subject is ≥ 12 years old.
* Subject is in good general health, based on medical history and vital signs.
* Subject is matched to the patient group for age, sex and BMI.

Exclusion Criteria:

Patients with ADPKD

* Subject has eczema, scleroderma, psoriasis, dermatitis, or any other abnormality on the skin of the dominant hand and/or lower back which, in the investigator's opinion, might interfere with the study assessments.
* Subject is currently undergoing dialysis, had a kidney transplant or is a user of tolvaptan.
* Female who is pregnant or breastfeeding.
* Simultaneous participation in another study which, in the investigator's opinion, might confound the results of the study.
* Subject is unable to refrain from drinking alcohol 24 hours prior to each study visit, and/or consumes ≥ 3 alcoholic consumptions per day.
* Subject is a regular user of cannabis, any illicit drugs and/or has a history of drug abuse.
* Subject is unable to refrain from drinking caffeinated beverages (such as coffee, tea, cola,…) 24 hours prior to each study visit.
* Subject has used concomitant drugs and/or treatments in a period smaller than or equal to 5 half-lives prior to enrollment, that may interfere, in the investigator's opinion, with the study results.
* Subject has a history of any illness or condition which, in the investigator's opinion, may interfere with safe and optimal participation in the study.

Healthy volunteers

* Subject has a history of any illness or condition which may affect the normal somatosensory functionality.
* Subject has eczema, scleroderma, psoriasis, dermatitis, or any other abnormality on the skin of the dominant hand and/or lower back which, in the investigator's opinion, might interfere with the study assessments.
* Female who is pregnant or breast-feeding.
* Simultaneous participation in another study which, in the investigator's opinion, might confound the results of the study.
* Subject is unable to refrain from drinking alcohol 24 hours prior to each study visit, and/or consumes ≥ 3 alcoholic consumptions per day.
* Subject is a regular user of cannabis, any illicit drugs and/or has a history of drug abuse.
* Subject is unable to refrain from drinking caffeinated beverages (such as coffee, tea, cola,…) 24 hours prior to each study visit.
* Subject has used concomitant drugs and/or treatments in a period smaller than or equal to 5 half-lives prior to enrollment, that may interfere, in the investigator's opinion, with the study results.
* Subject has a history of any illness or condition which, in the investigator's opinion, may interfere with safe and optimal participation in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ADPKD from the University Hospitals Leuven will be included in this study. Additionally, healthy volunteers will be included using the registered database of the Center for Clinical Pharmacology (UZ Leuven).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Somatosensory phenotyping of ADPKD using Quantitative Sensory Testing (QST) | Interval of ≤ 3 months between screening and study visit
  The somatosensory phenotype of patients with ADPKD will be evaluated using QST on the dominant hand and lower back. These results will be compared with the somatosensory phenotype of matched healthy volunteers.
Describing pain in ADPKD using the ADPKD-PDS questionnaire | Interval of ≤ 3 months between screening and study visit
  (Potential) pain in the last 7 days will be assessed using the ADPKD-PDS questionnaire, which contains 20 questions (1-5 Likert scale) in 7 domains: Dull Pain Severity, Sharp Pain Severity, Discomfort Severity, Overall Pain and Discomfort Severity, Dull Pain Interference, Sharp Pain Interference, and Discomfort Interference.
  Unit of Measure: Total score per domain
Describing neuropathic pain in ADPKD using the DN4 questionnaire | Interval of ≤ 3 months between screening and study visit
  The DN4 questionnaire will be used to evaluate whether the (potential) pain is neuropathic. The questionnaire consists of 10 yes/no questions, in which a total score of 4/10 or higher is considered indicative of neuropathic pain.
  Unit of Measure: Total DN4 score (/10)
Describing quality of life in ADPKD using the ADPKD-IS questionnaire | Interval of ≤ 3 months between screening and study visit
  Quality of life will be assessed using the ADPKD-IS questionnaire, which consists of 18 questions (1-5 Likert scale) in 3 domains (physical, emotional, fatigue) and 4 additional elements (guilt, sleep, size/shape of abdomen, urinary frequency/urgency).
  Unit of Measure: Total score per domain/element
Comparing pain between patients with ADPKD and healthy volunteers using the BPI-SF questionnaire | Interval of ≤ 3 months between screening and study visit
  The BPI-SF questionnaire consists of 9 questions, concerning both the intensity and impact of pain on daily functioning in the last 24 hours. This questionnaire will be conducted in patients with ADPKD and healthy volunteers.

SECONDARY OUTCOMES:
Correlation between QST and questionnaires | Interval of ≤ 3 months between screening and study visit
  A correlation between QST results and results from the questionnaires will be assessed in patients with ADPKD.
Differences in somatosensory phenotype depending on the disease stage of ADPKD | Interval of ≤ 3 months between screening and study visit
  Potential differences in somatosensory phenotype depending on the disease stage of patients with ADPKD (stage 1-5) will be evaluated using statistical analyses.
Differences in somatosensory phenotype depending on the sex of patients with ADPKD | Interval of ≤ 3 months between screening and study visit
  Potential differences in the somatosensory phenotype (QST) of female and male patients with ADPKD will be evaluated using statistical analyses.
Differences in pain and quality of life depending on the sex of patients with ADPKD | Interval of ≤ 3 months between screening and study visit
  Potential differences in pain and quality of life, described using questionnaires, of female and male patients with ADPKD will be evaluated using statistical analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Jan de Hoon, MD, PhD, MSc, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No